CLINICAL TRIAL: NCT03770494
Title: A Phase 1a/1b Study of LY3405105 Administered to Patients With Advanced Solid Tumors
Brief Title: A Study of LY3405105 in Participants With Advanced Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated for lack of sufficient efficacy.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17125; J1F-MC-JZFA (Other: Eli Lilly and Company); 2018-002668-23 (EudraCT Number)
Record Dates: First submitted 2018-12-07; First posted 2018-12-10 (Actual); Results first posted 2025-11-04 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LY3405105 (Experimental): This study was designed to be conducted in two phases:
  Phase 1a: This is a dose-escalation phase with a starting dose of LY3405105 1 milligram (mg) once daily (Part A1) or 2 mg three times per week (Part A2) on a 28-day cycle until confirmed progressive disease, unacceptable toxicity, or discontinuation for any other reason. Each dose-level will be determined and will have participants enrolled to it based on dose-limiting toxicity rate observed at previous dose-level. Intermediate, alternate, or higher dose levels will be explored if deemed necessary.
  Phase 1b: This is a dose-expansion phase designed to explore the anti-tumor activity of recommended LY3405105 dose and dosing schedule determined in phase 1a, in participants with multiple tumor types.
  [Phase 1b was planned but not initiated based on the sponsor's decision and limited efficacy observed in phase 1a]
  Interventions: Drug: LY3405105

INTERVENTIONS:
Drug: LY3405105 — Administered orally.

SUMMARY:
The main purpose of this study is to investigate the safety of LY3405105 in participants with advanced cancer. The study has two parts phase 1a and phase 1b. Participants will only enroll in one part.

ELIGIBILITY:
Inclusion Criteria:

Phase 1 a:

* Have histological or cytological evidence of a diagnosis of a solid tumor cancer that is advanced and/or metastatic
* Have available archived tissue for exploratory biomarker analysis
* Have adequate organ function
* Have discontinued all previous treatments for cancer and recovered from their side effects
* Are able to swallow capsules/tablets

Phase 1 b:

* Cohort 1: Triple-negative breast cancer (TNBC).
* Cohort 2: Clear cell ovarian cancer, endometrioid ovarian cancer, or endometrioid endometrial carcinoma with a LOF mutation in one or more of the following genes: ARID1A, KMT2C (MLL3), KMT2D (MLL2), or KDM6A (UTX).
* Cohort 3: Soft tissue sarcoma or sarcomatoid/rhabdoid malignancy with loss of expression of INI1, BRG1, or BRM by immunohistochemistry or a LOF mutation in one or more of the following genes: ARID1A, SMARCA2, SMARCA4, or SMARCB1. Participants aged ≥ 12 years with a body weight of ≥ 40 kilogram (kg) are acceptable for Cohorts 3. Participants with synovial sarcoma and a confirmed SS18-SSX gene fusion are also eligible.
* Cohort 4: Epithelioid sarcoma with INI1 loss of expression by immunohistochemistry or SMARCB1 LOF mutation. Participants aged ≥ 12 years with a body weight of ≥ 40 kilogram (kg) are acceptable for Cohorts 4.
* Cohort 5: Bladder cancer with a LOF mutation in one or more of the following genes: ARID1A, KMT2C (MLL3), KMT2D (MLL2), or KDM6A (UTX).

Exclusion Criteria:

* Have symptomatic central nervous system (CNS) malignancy or metastasis
* Have symptomatic human immunodeficiency virus (HIV), Hepatitis A, B, or C
* Have congestive heart failure
* Are breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2021-02-04 (Actual); Study Completion 2021-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (17):
- United States (7):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Smilow Cancer Hospital at Yale-New Haven, New Haven, Connecticut
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Pennsylvania Hospital, Philadelphia, Pennsylvania
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Princess Margaret Hospital, Toronto, Ontario, Canada
- France (3):
  - Institut Bergonie, Bordeaux
  - Institut Curie, Paris
  - Gustave Roussy, Villejuif
- Spain (2):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Madrid Norte Sanchinarro, Madrid
- Taiwan (4):
  - Taichung Veterans General Hospital, Taichung
  - National Cheng-Kung Uni. Hosp., Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garralda E, Schram AM, Bedard PL, Schwartz GK, Yuen E, McNeely SC, Ribeiro S, Cunningham J, Wang Y, Urunuela A, Xu X, LoRusso P. A Phase I Dose-Escalation Study of LY3405105, a Covalent Inhibitor of Cyclin-Dependent Kinase 7, Administered to Patients With Advanced Solid Tumors. Oncologist. 2024 Jan 5;29(1):e131-e140. doi: 10.1093/oncolo/oyad215. PMID 37531083
- [Derived] Sava GP, Fan H, Coombes RC, Buluwela L, Ali S. CDK7 inhibitors as anticancer drugs. Cancer Metastasis Rev. 2020 Sep;39(3):805-823. doi: 10.1007/s10555-020-09885-8. PMID 32385714
- See also: A Study of LY3405105 in Participants With Advanced Cancer — https://trials.lillytrialguide.com/en-US/trial/ISkx1UpFmMIUiQYaemQSE

RESULTS

PARTICIPANT FLOW:
Recruitment Details: * Phase 1a was a dose escalation phase with a starting dose of LY3405105 1 milligram (mg) once daily (Part A1) or 2 mg three times per week (Part A2) on a 28-day cycle until confirmed progressive disease, unacceptable toxicity, or discontinuation for any other reason. Each dose level will have minimum of 3 participants enrolled.
  * Phase 1b was a dose expansion phase which was planned but not initiated based on sponsor's decision and limited efficacy observed in phase 1a. No participants enrolled.
Pre-assignment Details: Completers included participants who died from any cause.
Groups:
- Part A1 Cohort 1 (1 mg, QD): Participants received 1 mg LY3405105 once daily (QD) orally on a 28-day cycle until confirmed progressive disease, unacceptable toxicity, or discontinuation for any other reason.
- Part A1 Cohort 2 (2 mg, QD): Participants received 2 mg LY3405105 QD orally on a 28-day cycle until confirmed progressive disease, unacceptable toxicity, or discontinuation for any other reason.
- Part A1 Cohort 3 (4 mg, QD): Participants received 3 mg LY3405105 QD orally on a 28-day cycle until confirmed progressive disease, unacceptable toxicity, or discontinuation for any other reason.
- Part A1 Cohort 4 (8 mg, QD): Participants received 8 mg LY3405105 QD orally on a 28-day cycle until confirmed progressive disease, unacceptable toxicity, or discontinuation for any other reason.
- Part A1 Cohort 5 (15 mg, QD): Participants received 15 mg LY3405105 QD orally on a 28-day cycle until confirmed progressive disease, unacceptable toxicity, or discontinuation for any other reason.
- Part A1 Cohort 6 (30 mg, QD): Participants received 30 mg LY3405105 QD orally on a 28-day cycle until confirmed progressive disease, unacceptable toxicity, or discontinuation for any other reason.
- Part A1 Cohort 7 (45 mg, QD): Participants received 45 mg LY3405105 QD orally on a 28-day cycle until confirmed progressive disease, unacceptable toxicity, or discontinuation for any other reason.
- Part A1 Cohort 8 (35 mg, QD): Participants received 35 mg LY3405105 QD orally on a 28-day cycle until confirmed progressive disease, unacceptable toxicity, or discontinuation for any other reason.
- Part A1 Cohort 9 (25 mg, QD): Participants received 25 mg LY3405105 QD orally on a 28-day cycle until confirmed progressive disease, unacceptable toxicity, or discontinuation for any other reason.
- Part A1 Cohort 10 (20 mg, QD): Participants received 20 mg LY3405105 QD orally on a 28-day cycle until confirmed progressive disease, unacceptable toxicity, or discontinuation for any other reason.
- Part A2 Cohort 1 (2 mg, TIW): Participants received 2 mg LY3405105 three times per week (TIW) orally on a 28-day cycle until confirmed progressive disease, unacceptable toxicity, or discontinuation for any other reason.
- Part A2 Cohort 2 (4 mg, TIW): Participants received 4 mg LY3405105 TIW orally on a 28-day cycle until confirmed progressive disease, unacceptable toxicity, or discontinuation for any other reason.
- Part A2 Cohort 3 (8 mg, TIW): Participants received 8 mg LY3405105 TIW orally on a 28-day cycle until confirmed progressive disease, unacceptable toxicity, or discontinuation for any other reason.
- Phase 1b: This is a dose-expansion phase designed to explore the anti-tumor activity of recommended LY3405105 dose and dosing schedule determined in phase 1a, in participants with multiple tumor types.
Period: Overall Study
Arm/Group | Part A1 Cohort 1 (1 mg, QD) | Part A1 Cohort 2 (2 mg, QD) | Part A1 Cohort 3 (4 mg, QD) | Part A1 Cohort 4 (8 mg, QD) | Part A1 Cohort 5 (15 mg, QD) | Part A1 Cohort 6 (30 mg, QD) | Part A1 Cohort 7 (45 mg, QD) | Part A1 Cohort 8 (35 mg, QD) | Part A1 Cohort 9 (25 mg, QD) | Part A1 Cohort 10 (20 mg, QD) | Part A2 Cohort 1 (2 mg, TIW) | Part A2 Cohort 2 (4 mg, TIW) | Part A2 Cohort 3 (8 mg, TIW) | Phase 1b
Started | 4 | 4 | 4 | 4 | 5 | 5 | 5 | 3 | 3 | 6 | 4 | 4 | 3 | 0
Received At Least 1 Dose of Study Drug | 4 | 4 | 4 | 4 | 5 | 5 | 5 | 3 | 3 | 6 | 4 | 4 | 3 | 0
Completed | 2 | 1 | 2 | 2 | 1 | 1 | 2 | 1 | 0 | 1 | 2 | 2 | 3 | 0
Not Completed | 2 | 3 | 2 | 2 | 4 | 4 | 3 | 2 | 3 | 5 | 2 | 2 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Study terminated by sponsor | 1 | 2 | 1 | 1 | 1 | 2 | 1 | 2 | 1 | 2 | 1 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 2 | 2 | 2 | 0 | 2 | 3 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants. Only phase 1a participants baseline characters reported as no participant enrolled in phase 1b.
Groups:
- Part A2 Cohort 1 (2 mg, TIW): Participants received 2 mg LY3405105 TIW orally on a 28-day cycle until confirmed progressive disease, unacceptable toxicity, or discontinuation for any other reason.
- Total: Total of all reporting groups
Arm/Group | Part A1 Cohort 1 (1 mg, QD) | Part A1 Cohort 2 (2 mg, QD) | Part A1 Cohort 3 (4 mg, QD) | Part A1 Cohort 4 (8 mg, QD) | Part A1 Cohort 5 (15 mg, QD) | Part A1 Cohort 6 (30 mg, QD) | Part A1 Cohort 7 (45 mg, QD) | Part A1 Cohort 8 (35 mg, QD) | Part A1 Cohort 9 (25 mg, QD) | Part A1 Cohort 10 (20 mg, QD) | Part A2 Cohort 1 (2 mg, TIW) | Part A2 Cohort 2 (4 mg, TIW) | Part A2 Cohort 3 (8 mg, TIW) | Total
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 5 | 5 | 5 | 3 | 3 | 6 | 4 | 4 | 3 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 1 | 3 | 2 | 2 | 4 | 0 | 3 | 4 | 3 | 3 | 2 | 32
  >=65 years | 1 | 2 | 3 | 1 | 3 | 3 | 1 | 3 | 0 | 2 | 1 | 1 | 1 | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 2 | 3 | 4 | 2 | 5 | 2 | 3 | 5 | 3 | 4 | 1 | 41
  Male | 1 | 0 | 2 | 1 | 1 | 3 | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 4
  White | 3 | 3 | 3 | 4 | 4 | 5 | 4 | 2 | 1 | 5 | 4 | 3 | 2 | 43
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 7
  Spain | 3 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 1 | 4 | 2 | 1 | 17
  United States | 1 | 2 | 3 | 2 | 3 | 4 | 3 | 1 | 2 | 5 | 0 | 2 | 2 | 30

OUTCOME MEASURES:

1. Primary Outcome: Phase 1a: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: A DLT is a clinically significant adverse event that is possibly related to the study drug and fulfils any one of the following criteria using the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) v4.0:
  1) Nonhematologic Grade ≥3 toxicity, except nausea, constipation, diarrhoea, vomiting or electrolyte disturbance lasting for <72 hours and can be controlled with treatment, fatigue/anorexia lasting for <5 days, transient grade 3 elevations of alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST), without evidence of other hepatic injury; 2) Total bilirubin >2×upper limit of normal (ULN) with ALT/AST >3×ULN in the absence of cholestasis (alkaline phosphatase <2×ULN); 3) Grade 4 neutropenia >5 days duration, Any febrile neutropenia, Grade 4 thrombocytopenia of any duration, Grade 3 thrombocytopenia with clinically significant bleeding, Grade 3/4 anemia or any other significant toxicity deemed to be dose limiting by investigators.
Time Frame: Cycle 1 (Up To 28 Days)
Population: All phase 1a participants who received at least one dose of LY3405105 in Cycle 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A1 Cohort 1 (1 mg, QD) | Part A1 Cohort 2 (2 mg, QD) | Part A1 Cohort 3 (4 mg, QD) | Part A1 Cohort 4 (8 mg, QD) | Part A1 Cohort 5 (15 mg, QD) | Part A1 Cohort 6 (30 mg, QD) | Part A1 Cohort 7 (45 mg, QD) | Part A1 Cohort 8 (35 mg, QD) | Part A1 Cohort 9 (25 mg, QD) | Part A1 Cohort 10 (20 mg, QD) | Part A2 Cohort 1 (2 mg, TIW) | Part A2 Cohort 2 (4 mg, TIW) | Part A2 Cohort 3 (8 mg, TIW)
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 5 | 5 | 5 | 3 | 3 | 6 | 4 | 4 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 1 | 0 | 0 | 0 | 0

2. Secondary Outcome: Phase 1a (Part A1): Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Time Zero to 24 Hours [AUC(0-24)] of LY3405105
Description: AUC(0-24) of LY3405105
Time Frame: Cycle 1 Day 1 (Predose, 1, 2, 4, 6, 8, 24 hours post-dose)
Population: All part A1 participants of phase 1a who received at least one dose of LY3405105 and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours per milliliter (ng*h/mL)
Arm/Group | Part A1 Cohort 1 (1 mg, QD) | Part A1 Cohort 2 (2 mg, QD) | Part A1 Cohort 3 (4 mg, QD) | Part A1 Cohort 4 (8 mg, QD) | Part A1 Cohort 5 (15 mg, QD) | Part A1 Cohort 6 (30 mg, QD) | Part A1 Cohort 7 (45 mg, QD) | Part A1 Cohort 8 (35 mg, QD) | Part A1 Cohort 9 (25 mg, QD) | Part A1 Cohort 10 (20 mg, QD)
Number analyzed (Participants) | 4 | 4 | 3 | 4 | 5 | 4 | 5 | 1 | 1 | 4
nanograms*hours per milliliter (ng*h/mL) | 12.1 (63) | 30.3 (140) | 91.3 (120) | 102 (24) | 159 (148) | 775 (24) | 1730 (104) | NA (NA) — N=1, Geometric mean and coefficient of variation were not calculated. Individual value reported: 623 ng*h/mL. | NA (NA) — N=1, Geometric mean and coefficient of variation were not calculated. Individual value reported: 599 ng*h/mL. | 328 (80)

3. Secondary Outcome: Phase 1a (Part A1): PK: Area Under the Concentration Versus Time Curve During One Dosing Interval [AUC(Tau)] of LY3405105
Description: AUC of LY3405105 during one dosing interval of 24 hours [tau = 24 hours].
Time Frame: Cycle 1 Day 15 (Predose, 1, 2, 4, 6, 8, 24 hours post-dose)
Population: All part A1 participants of phase 1a who received at least one dose of LY3405105 and had evaluable PK data. For Part A1 Cohort 7 (45 mg, QD) and Cohort 9 (25 mg, QD), day 15 PK data was not collected for any participants as study was terminated prior to data collection; thus, zero participants were analysed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part A1 Cohort 1 (1 mg, QD) | Part A1 Cohort 2 (2 mg, QD) | Part A1 Cohort 3 (4 mg, QD) | Part A1 Cohort 4 (8 mg, QD) | Part A1 Cohort 5 (15 mg, QD) | Part A1 Cohort 6 (30 mg, QD) | Part A1 Cohort 7 (45 mg, QD) | Part A1 Cohort 8 (35 mg, QD) | Part A1 Cohort 9 (25 mg, QD) | Part A1 Cohort 10 (20 mg, QD)
Number analyzed (Participants) | 4 | 4 | 3 | 4 | 3 | 4 | 0 | 2 | 0 | 4
ng*h/mL | 22.6 (37) | 47.4 (115) | 132 (74) | 153 (46) | 208 (25) | 1620 (53) |  | NA (NA) — N=2, Geometric mean and coefficient of variation were not calculated. Individual values reported: 1760 ng*h/mL, 3610 ng*h/mL |  | NA (NA) — Due to insufficient quantifiable data, AUC(Tau) couldn't be calculated for any of the participants.

4. Secondary Outcome: Phase 1a (Part A2): PK: Area Under the Concentration Versus Time Curve From Time Zero to Infinity [AUC(0-∞)] of LY3405105
Description: AUC(0-∞) of LY3405105.
Time Frame: Cycle 1 Day 1 (Predose, 1, 2, 4, 6, 8, 24, 48 hours post-dose)
Population: All part A2 participants of phase 1a who received at least one dose of LY3405105 and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part A2 Cohort 1 (2 mg, TIW) | Part A2 Cohort 2 (4 mg, TIW) | Part A2 Cohort 3 (8 mg, TIW)
Number analyzed (Participants) | 3 | 3 | 2
ng*h/mL | 43.5 (88) | 63.3 (48) | NA (NA) — N=2, Geometric mean and coefficient of variation were not calculated. Individual values reported: 73.9 ng*h/mL, 113 ng*h/mL

5. Secondary Outcome: Phase 1a (Part A2): PK: Area Under the Concentration Versus Time Curve During One Dosing Interval [AUC(Tau)] of LY3405105
Description: AUC of LY3405105 during one dosing interval of 48 hours [tau = 48 hours].
Time Frame: Cycle 1 Day 15 (Predose, 1, 2, 4, 6, 8, 24, 48 hours post-dose)
Population: All part A2 participants of phase 1a who received at least one dose of LY3405105 and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part A2 Cohort 1 (2 mg, TIW) | Part A2 Cohort 2 (4 mg, TIW) | Part A2 Cohort 3 (8 mg, TIW)
Number analyzed (Participants) | 4 | 3 | 3
ng*h/mL | 70.5 (81) | 32.6 (201) | 163 (25)

6. Secondary Outcome: Phase 1a: Objective Response Rate (ORR): Percentage of Participants With a Confirmed Complete Response (CR) or Partial Response (PR)
Description: ORR is the best overall tumor response of complete response (CR) or partial response (PR) as classified by the investigator according to the Response Evaluation Criteria In Solid Tumors (RECIST v1.1). CR is defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR is defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions.
Time Frame: Baseline through Measured Progressive Disease (Up To 349 Days)
Population: All phase 1a participants who received at least one dose of LY3405105.
Measure: Number; unit: Percentage of participants
Arm/Group | Part A1 Cohort 1 (1 mg, QD) | Part A1 Cohort 2 (2 mg, QD) | Part A1 Cohort 3 (4 mg, QD) | Part A1 Cohort 4 (8 mg, QD) | Part A1 Cohort 5 (15 mg, QD) | Part A1 Cohort 6 (30 mg, QD) | Part A1 Cohort 7 (45 mg, QD) | Part A1 Cohort 8 (35 mg, QD) | Part A1 Cohort 9 (25 mg, QD) | Part A1 Cohort 10 (20 mg, QD) | Part A2 Cohort 1 (2 mg, TIW) | Part A2 Cohort 2 (4 mg, TIW) | Part A2 Cohort 3 (8 mg, TIW)
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 5 | 5 | 5 | 3 | 3 | 6 | 4 | 4 | 3
Percentage of participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Phase 1a: Disease Control Rate (DCR): Percentage of Participants Who Exhibit Stable Disease (SD), Confirmed CR or PR
Description: DCR is the percentage of participants with a best overall response of CR, PR or SD as defined by RECIST v1.1. CR is defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR is defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions. SD is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD) for target lesions, no progression of non-target lesions, and no appearance of new lesions. PD is defined as at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions.
Time Frame: Baseline through Measured Progressive Disease (Up To 349 Days)
Population: All phase 1a participants who received at least one dose of LY3405105.
Measure: Number; unit: Percentage of participants
Arm/Group | Part A1 Cohort 1 (1 mg, QD) | Part A1 Cohort 2 (2 mg, QD) | Part A1 Cohort 3 (4 mg, QD) | Part A1 Cohort 4 (8 mg, QD) | Part A1 Cohort 5 (15 mg, QD) | Part A1 Cohort 6 (30 mg, QD) | Part A1 Cohort 7 (45 mg, QD) | Part A1 Cohort 8 (35 mg, QD) | Part A1 Cohort 9 (25 mg, QD) | Part A1 Cohort 10 (20 mg, QD) | Part A2 Cohort 1 (2 mg, TIW) | Part A2 Cohort 2 (4 mg, TIW) | Part A2 Cohort 3 (8 mg, TIW)
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 5 | 5 | 5 | 3 | 3 | 6 | 4 | 4 | 3
Percentage of participants | 75 | 50 | 0 | 0 | 20 | 40 | 20 | 66.7 | 33.3 | 0 | 50 | 75 | 0

8. Secondary Outcome: Phase 1a: Duration of Response (DOR)
Description: DoR will be calculated only for responders. It is measured from the date of first evidence of a confirmed CR or PR response to the date of first progression of disease or the date of death due to any cause, whichever is earlier.
Time Frame: Date of Confirmed CR or PR to Date of Objective Progression or Death Due to Any Cause (Estimated up to 12 Months)
Population: Zero participants analysed. DoR was not evaluable as there were no participants with CR or PR.
Arm/Group | Part A1 Cohort 1 (1 mg, QD) | Part A1 Cohort 2 (2 mg, QD) | Part A1 Cohort 3 (4 mg, QD) | Part A1 Cohort 4 (8 mg, QD) | Part A1 Cohort 5 (15 mg, QD) | Part A1 Cohort 6 (30 mg, QD) | Part A1 Cohort 7 (45 mg, QD) | Part A1 Cohort 8 (35 mg, QD) | Part A1 Cohort 9 (25 mg, QD) | Part A1 Cohort 10 (20 mg, QD) | Part A2 Cohort 1 (2 mg, TIW) | Part A2 Cohort 2 (4 mg, TIW) | Part A2 Cohort 3 (8 mg, TIW)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Phase 1a: Time to Response (TTR)
Description: TTR is defined as the time from the date of start of treatment to the date measurement criteria for confirmed CR or PR (whichever is first recorded) are first met.
Time Frame: Baseline to Date of Confirmed CR or PR (Estimated up to 6 Months)
Population: Zero participants analysed. TTR was not evaluable as there were no participants with CR or PR.
Arm/Group | Part A1 Cohort 1 (1 mg, QD) | Part A1 Cohort 2 (2 mg, QD) | Part A1 Cohort 3 (4 mg, QD) | Part A1 Cohort 4 (8 mg, QD) | Part A1 Cohort 5 (15 mg, QD) | Part A1 Cohort 6 (30 mg, QD) | Part A1 Cohort 7 (45 mg, QD) | Part A1 Cohort 8 (35 mg, QD) | Part A1 Cohort 9 (25 mg, QD) | Part A1 Cohort 10 (20 mg, QD) | Part A2 Cohort 1 (2 mg, TIW) | Part A2 Cohort 2 (4 mg, TIW) | Part A2 Cohort 3 (8 mg, TIW)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Phase 1b: Progression Free Survival (PFS)
Description: PFS is defined as the time from the date of start of treatment to the first date of radiologically documented progressive disease or the date of death due to any cause, whichever occurs first.
Time Frame: Baseline to Objective Progression or Death Due to Any Cause (Estimated up to 12 Months)
Population: PFS is a phase 1b outcome measure. Phase 1b of the study is not conducted and no participant enrolled, thus no data collected.
Arm/Group | Phase 1b
Number analyzed (Participants) | 0

11. Secondary Outcome: Phase 1b: Overall Survival (OS)
Description: OS is defined as the time from the date of start of treatment to the date of death due to any cause.
Time Frame: Baseline to Date of Death from Any Cause (Estimated up to 12 Months)
Population: OS is a phase 1b outcome measure. Phase 1b of the study is not conducted and no participant enrolled, thus no data collected.
Arm/Group | Phase 1b
Number analyzed (Participants) | 0

12. Primary Outcome: Phase 1b: Objective Response Rate (ORR): Percentage of Participants With a Confirmed Complete Response (CR) or Partial Response (PR)
Description: as for outcome 6
Time Frame: Baseline through Measured Progressive Disease (Estimated up to 6 Months)
Population: ORR is phase 1b primary outcome measure. Phase 1b of the study is not conducted and no participant enrolled, thus no data collected.
Arm/Group | Phase 1b
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Baseline to Follow-up (Up To 690 Days)
Description: All phase 1a participants who received at least one dose of LY3405105. Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly.
Arm/Group | Part A1 Cohort 1 (1 mg, QD) | Part A1 Cohort 2 (2 mg, QD) | Part A1 Cohort 3 (4 mg, QD) | Part A1 Cohort 4 (8 mg, QD) | Part A1 Cohort 5 (15 mg, QD) | Part A1 Cohort 6 (30 mg, QD) | Part A1 Cohort 7 (45 mg, QD) | Part A1 Cohort 8 (35 mg, QD) | Part A1 Cohort 9 (25 mg, QD) | Part A1 Cohort 10 (20 mg, QD) | Part A2 Cohort 1 (2 mg, TIW) | Part A2 Cohort 2 (4 mg, TIW) | Part A2 Cohort 3 (8 mg, TIW)
All-Cause Mortality (participants affected / at risk) | 2/4 | 1/4 | 2/4 | 2/4 | 1/5 | 1/5 | 2/5 | 1/3 | 0/3 | 1/6 | 2/4 | 3/4 | 3/3
Serious Adverse Events (participants affected / at risk) | 2/4 | 1/4 | 0/4 | 0/4 | 0/5 | 1/5 | 2/5 | 3/3 | 1/3 | 1/6 | 2/4 | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 4/4 | 4/4 | 4/5 | 5/5 | 5/5 | 3/3 | 3/3 | 6/6 | 3/4 | 4/4 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A1 Cohort 1 (1 mg, QD) (N=4) | Part A1 Cohort 2 (2 mg, QD) (N=4) | Part A1 Cohort 3 (4 mg, QD) (N=4) | Part A1 Cohort 4 (8 mg, QD) (N=4) | Part A1 Cohort 5 (15 mg, QD) (N=5) | Part A1 Cohort 6 (30 mg, QD) (N=5) | Part A1 Cohort 7 (45 mg, QD) (N=5) | Part A1 Cohort 8 (35 mg, QD) (N=3) | Part A1 Cohort 9 (25 mg, QD) (N=3) | Part A1 Cohort 10 (20 mg, QD) (N=6) | Part A2 Cohort 1 (2 mg, TIW) (N=4) | Part A2 Cohort 2 (4 mg, TIW) (N=4) | Part A2 Cohort 3 (8 mg, TIW) (N=3)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronavirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ophthalmic herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Part A1 Cohort 1 (1 mg, QD) (N=4) | Part A1 Cohort 2 (2 mg, QD) (N=4) | Part A1 Cohort 3 (4 mg, QD) (N=4) | Part A1 Cohort 4 (8 mg, QD) (N=4) | Part A1 Cohort 5 (15 mg, QD) (N=5) | Part A1 Cohort 6 (30 mg, QD) (N=5) | Part A1 Cohort 7 (45 mg, QD) (N=5) | Part A1 Cohort 8 (35 mg, QD) (N=3) | Part A1 Cohort 9 (25 mg, QD) (N=3) | Part A1 Cohort 10 (20 mg, QD) (N=6) | Part A2 Cohort 1 (2 mg, TIW) (N=4) | Part A2 Cohort 2 (4 mg, TIW) (N=4) | Part A2 Cohort 3 (8 mg, TIW) (N=3)
Anaemia (Blood and lymphatic system disorders) | 3 (7) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (6) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (4) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periorbital oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 2 (4) | 2 (3) | 1 (1) | 1 (1) | 1 (1) | 2 (3)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (7) | 1 (1) | 1 (1) | 1 (1) | 4 (9) | 4 (5) | 3 (11) | 2 (2) | 3 (4) | 0 (0) | 2 (2) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 3 (4) | 1 (1) | 2 (3) | 1 (2) | 3 (3) | 0 (0) | 3 (3) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 2 (7) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (2) | 2 (3) | 1 (1) | 1 (2) | 3 (3) | 2 (3) | 1 (8) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary tract infection (Infections and infestations) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ophthalmic herpes zoster (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (3) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0/3 (0) | 1 (1) | 0/2 (0) | 0/3 (0) | 0/4 (0) | 0/2 (0) | 0 (0) | 0/2 (0) | 0 (0) | 0/5 (0) | 0/3 (0) | 0 (0) | 0/1 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 2 (5) | 1 (1) | 1 (1) | 1 (3) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 2 (5) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Blood alkaline phosphatase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Electrocardiogram qt prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (6) | 2 (7) | 3 (11) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Troponin i increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 2 (4) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nystagmus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chromaturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-08-13): https://cdn.clinicaltrials.gov/large-docs/94/NCT03770494/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-20): https://cdn.clinicaltrials.gov/large-docs/94/NCT03770494/SAP_001.pdf